CLINICAL TRIAL: NCT02115126
Title: A Randomized Phase II Trial to Evaluate an EBV Derived Dendritic Cell (DC) Vaccine When Administered Alone or Co-administered With the TLR9 Agonist, DUK-CPG-001, in EBV+ Lymphoma in the Setting of Autologous Stem Cell Transplant
Brief Title: Phase II Trial to Evaluate an EBV-derived Dendritic Cell Vaccine in Autologous Stem Cell Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00042574
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Hodgkin Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMP2A-loaded conventional DC vaccine (Active Comparator): Epstein-Barr virus (EBV) derived tumor antigen, LMP2 loaded DC vaccine
  Interventions: Biological: LMP2A-loaded conventional DC vaccine
- LMP2A-loaded DC vaccine + DUK-CPG-001 (Experimental): Epstein-Barr virus (EBV) derived tumor antigen, LMP2 loaded DC vaccine co-administered with a Toll-like receptor 9 (TLR9) ligand, DUK-CPG-001
  Interventions: Biological: DUK-CPG-001

INTERVENTIONS:
Biological: LMP2A-loaded conventional DC vaccine — Vaccine #1 will be administered 9-13 weeks status post peripheral blood stem cell (PBSC) infusion. At the time of vaccination, ANC must be > 1.5.
  Vaccine #2, the booster vaccine, will be administered 4 weeks +/- 7 days status post vaccine #1. At the time of vaccination, ANC must be > 1.5.
  Vaccines will be administered following standard institutional practice for IV infusions using a peripheral or central line and following sterile technique. On the day of vaccination, the patient will be given a total dose of 3 x 107 cells in 30ml of normal saline per vaccination.
  Arms: LMP2A-loaded conventional DC vaccine
Biological: DUK-CPG-001 — On the day of vaccination, for those patients who are randomized to receive DUK-CPG-001, a single vial will be dispensed to the nurse, upon request, by Duke ICS. DUK-CPG-001 will be thawed at room temperature right before use and 0.5 ml (5 mg) will be injected subcutaneously immediately after vaccination.
  DUK-CPG-001 will be stored at -20ºC until use. It will be stored in the Duke Investigational Chemotherapy Service pharmacy.
  Using standard institutional guidelines and sterile technique for subcutaneous injections, 5 mg of DUK-CPG-001 will be injected subcutaneously immediately after each vaccination.
  Arms: LMP2A-loaded DC vaccine + DUK-CPG-001

SUMMARY:
This is a non-blinded, not placebo controlled, randomized, parallel phase 2 pilot study to evaluate the immunological response and the safety of Epstein Barr Virus (EBV)-derived tumor antigen, Latent Membrane Protein-2 (LMP2)-loaded dendritic cell (DC) vaccines alone or co-administered with the TLR9 ligand, DUK-CPG-001, in patients with EBV+ lymphoma in the setting of autologous stem cell transplant with infusion of mature T cells. Patients will be randomized to receive vaccine alone or vaccine co-administered with the TLR9 ligand, DUK-CPG-001. Randomization will be stratified by 2 disease types: Hodgkin lymphoma and non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
Objectives

The primary objectives of this study are to:

1. To assess the ability of an Epstein-Barr virus (EBV) derived tumor antigen, LMP2 loaded DC vaccine co-administered with a Toll-like receptor 9 (TLR9) ligand, DUK-CPG-001, to induce EBV derived tumor antigen specific CD8+ T cell response in patients with EBV+ lymphoma in the setting of autologous stem cell transplant
2. To assess the ability of an Epstein-Barr virus (EBV) derived tumor antigen, LMP2 loaded DC vaccine administered alone to induce EBV derived tumor antigen specific CD8+ T cell response in patients with EBV+ lymphoma in the setting of autologous stem cell transplant
3. To evaluate the safety of using LMP2- loaded DC vaccine alone or co-administered with the TLR9 ligand, DUK-CPG-001, in patients with EBV+ lymphoma in the setting of autologous stem cell transplant

The secondary objectives of this study are to:

1. Evaluate duration of the presence of long term memory cells after administration of an LMP2 loaded DC vaccine alone or co-administered with the TLR9 ligand, DUK-CPG-001.
2. Evaluate duration of multi-functional CD8 T cell responses after administration of an LMP2 loaded DC vaccine alone or co-administered with the TLR9 ligand, DUK-CPG-001.
3. Evaluate duration of Th1, Th2 and Th17 CD4 T cell responses as well as CD4+CD25+Foxp3+ regulatory T cell (Treg) responses after administration of an LMP2 loaded DC vaccine alone or co-administered with the TLR9 ligand, DUK-CPG-001.
4. Evaluate the disease free survival (DFS) of patients with EBV+ lymphoma in the setting of autologous stem cell transplant who receive LMP2-loaded DC vaccines alone or co-administered with DUK-CPG-001.

Patient population Patients with EBV+ lymphoma who are in a complete remission (CR) after salvage therapy with plans to proceed to autologous peripheral stem cell transplant .

Immune response will be defined as an increase in number of spots to 25-fold more than at baseline, or at least 200 spots per 105 CD8+ T cells, by Day 7 post 2nd vaccination (i.e., a patient with a baseline of 1 spot/105 CD8+ T cells who achieved 25 spots/million would not be counted as a response).

1. Leukapheresis #1: The first pheresis will be performed after that patient has obtained a complete remission, but prior to transplant. Complete remission will be determined based on Cheson Criteria100. No special preparative regimen is required prior to pheresis but it must occur at least 2 weeks after most recent chemotherapy and most recent granulocytic growth factor.

   Pheresis will last approximately 4 hours to collect a goal of 1 x 108 nucleated cells/kg. This will follow standard stem cell transplant Standard Operating Procedures (SOPs). The cells will be transferred to John Sampson's GMP facility (Duke Brain Tumor Immunotherapy Processing Laboratory) where the sample will be divided into DC cell product for making vaccine, T cells for re-infusion during transplant, and research sample that will go to Yiping Yang's lab.

   As described below, they will subsequently be defrosted and the T cells will be infused at the time of the autologous stem cell transplant. This will follow standard stem cell transplant Standard Operating Procedures (SOPs).Please see appendix 8.6 Cell collection: removal of PBMCs by leukapheresis.
2. Leukapheresis # 2: This is a standard-of-care pheresis to collect cells for the autologous stem cell transplant and will be performed as per the usual stem cell transplant and pheresis SOP.

   Leukapheresis will follow institutional norms.
3. Stem Cell Transplant will follow institutional norms. The standard minimum infusion of CD34+ PBSC cells required for autologous stem cell transplant is 2 x 106 cd34+ cells/kg (range 2-7). The standard transplant preparative regimens used are BEAM or BCV.
4. T Cell Infusion: T cells will be thawed and infused through an IV after the autologous stem cell graft infusion has been completed. This will be infused following the stem cell transplant Standard Operating Procedure (SOP) for re-infusion of thawed transplant products (SOP ABMT-GEN-017).
5. Post Transplant Vaccine #1: Nine -13 weeks status PBSC transplant, patients will receive their first post-transplant vaccination. At the time of vaccination, ANC must be > 1.5. Delays beyond 13 weeks may be allowed after discussion with the PI. Delays beyond the 13 weeks will be decided on by the PI on a case by case basis but will only be allowed if delay is due to a slow ANC recovery that has been attributed to a medication or if the delay was for a non-medical reason.
6. Post Transplant Vaccine #2: Four weeks +/- 7 days after post-transplant vaccine #1, a second Boost vaccination will be administered. At the time of vaccination ANC must be > 1.5.

1. Subjects who are randomized to the CPG arm will receive CPG immediately after vaccine #1 and vaccine #2.

7) Blood samples for evaluation of immune response will be collected throughout the study procedures. Specifically, blood samples will be obtained within 7 days prior to initial leukapheresis. Blood will also be collected prior to receiving vaccine # 1 and #2 on the day on which vaccine is administered or up to 2 days before hand. In addition, blood will be drawn 7 days after each vaccination and at one, three and six months after the second vaccination. These blood samples will be used for analyzing T cell responses as detailed in section 3.7. The day 7 draws must be drawn +/- 2 day. The one, three and six month draws may occur +/- 1 week.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria:

* Patient must have a histologically proven diagnosis of any EBV+ Hodgkin or non-Hodgkin lymphoma
* EBV positive will be defined as positive if LMP1 or 2 or EBER are positive. As long as EBV positive on a prior biopsy, EBV testing will not be required at the time of relapse. However, if EBV testing performed on a more recent biopsy and it is negative, that patient will be excluded.
* Patients must have had persistent, relapsed, or refractory disease to at least one prior regimen with plans to proceed to autologous stem cell transplant
* Patients must be in a complete remission at time of initial pheresis for vaccine preparation; complete remission will be determined using Cheson Criteria100
* There are no limits on the number of prior therapies allowed
* Able to give voluntary written informed consent
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study therapy and for 3 months after vaccine #2.
* Male subject agrees to use an acceptable method for contraception for the duration of the study therapy and for 3 months after vaccine #2.
* Patients must be 18 years of age or older.
* ECOG performance status 0-2.

Exclusion Criteria

* An estimated or measured creatinine clearance of less than 30 ml/min.
* AST, ALT, total bilirubin > 3 times the upper limit of normal
* Patients on chronic immunosuppressive therapy for any reason (other than chemotherapy for HL)
* Chronic systemic steroid therapy at doses greater than 10mg/day of prednisone or its equivalent.
* Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result within 48 hours of enrollment. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs for this disease within 14 days of enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients who are HIV positive AND have a CD4 count <50
* Prior solid organ transplant or allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2020-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Immune response | 7 days post 2nd vaccination
  Immune response will be defined as an increase in number of spots to 25-fold more than at baseline, and at least 200 spots per 105 cluster of differentiation 8 (CD8)+ T cells, by Day 7 post 2nd vaccination (i.e., a patient with a baseline of 1 spot/105 CD8+ T cells who achieved 25 spots/million would not be counted as a response).
  "Spots" are the readout for immune activation measured by the enzyme-linked immunosorbent spot (ELISPOT) assay. Each spot is indicative of an activated T cell that secrete interferon (IFN)-gamma, a cytokine produced by activated T cells.

SECONDARY OUTCOMES:
Number of patients with greater than grade 1 toxicity | 30 days post last dose of vaccine
Duration of the presence of long term memory cells | 7 days post second dose of vaccine
Duration of multi-functional CD8 T cell responses | 7 days post second dose of vaccine
Duration of Th1, Th2 and Th17 cluster of differentiation 4 (CD4) T cell responses as well as CD4+cluster of differentiation 25 (CD25)+Foxp3+ regulatory T cell (Treg) responses | 7 days post second dose of vaccine
Disease free survival | up to 10 years
  Number of days from PBSC transplant until disease relapse or death

CONTACTS AND LOCATIONS:
Overall Officials: Anne Beaven, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States